CLINICAL TRIAL: NCT06583551
Title: Comparison of the Effectiveness of Botox, Dry Needling, Pharmacological Treatment, and Manual Therapy for Bruxism-Induced Myalgia: a Prospective Randomized Study
Brief Title: Effectiveness of Botox, Dry Needling, Pharmacological Treatment, and Manual Therapy for Bruxism-Induced Myalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20/120
Record Dates: First submitted 2024-08-29; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2021-01

CONDITIONS: Myalgia; Bruxism; Quality of Life
Keywords: myalgia; Botulinum toxin; bruxism; Dry needling; manual therapy
MeSH Terms: conditions — Myalgia; Bruxism | interventions — Botulinum Toxins; incobotulinumtoxinA; Dry Needling; Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Group 1: Botulinum toxin (BTX-A) injection (n=20) Group 2: Dry needling (DN) (n=20) Group 3: Pharmacological therapy (PT) (n=20) Group 4: Manual therapy (MT) (n=20)
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were informed only about the type of treatment they received. The results were measured and recorded by another researcher other than the operator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Active Comparator): A single session of Botox (Botulinum toxin A) injection was performed. 50 IU was administered bilaterally by intramuscular injection: 30 IU within the masseter muscles and 20 IU within the anterior temporalis muscles.
  Interventions: Drug: Botulinum toxin
- Group 2 (Active Comparator): Dry needling was performed using sterile plastic cylindrical guide needles (25 mm length, 0.25 mm diameter) The needles were inserted 5 mm deep into hypertonic and irritable nodules (trigger points, TrPs) within the masseter and temporalis muscles. Each needle was rotated twice clockwise and then removed after remaining in the TrPs for a total of 20 minutes. The treatment was administered in three sessions, each one week apart.
  Interventions: Procedure: Dry needling
- Group 3 (Active Comparator): Pharmacological treatment was administered by prescribing Miyorel, a combination of methocarbamol (380 mg) and paracetamol (300 mg). The prescribed dosage was two tablets, taken three times daily, for a period of three weeks.
  Interventions: Drug: Myorel
- Group 4 (Active Comparator): Manual therapy was administered, consisting of bilateral facial massage and stretching maneuvers targeting the masseter and temporalis muscles. This treatment was performed for 20 minutes daily over a period of three weeks.
  Interventions: Procedure: Manual therapy

INTERVENTIONS:
Drug: Botulinum toxin — Botulinum toxin, produced by Clostridium botulinum, is a neurotoxin. Presently, there are 7 serotypes (A, B, C1, D, E, F, G). Botulinum neurotoxin A (BoNT-A) is the most frequently used variant in clinical applications.
  Other Names: Intramuscular injection of Botulinum toxin A. (BoNT-A)
  Arms: Group 1
Procedure: Dry needling — Dry needling (DN) is a type of acupuncture therapy, that uses a thin filiform needle to penetrate the skin and stimulate underlying myofascial trigger points (MTrPs) and muscular, and connective tissues.
  Arms: Group 2
Drug: Myorel — Metacarbamol (380mg), paracetamol (300mg)
  Arms: Group 3
Procedure: Manual therapy — Manual therapy (MT) entails the use of the hands to apply a force with a therapeutic intent, including techniques such as massage, joint mobilization/manipulation, myofascial release, nerve manipulation, strain/counterstrain, and acupressure.
  Arms: Group 4

SUMMARY:
Eighty individuals (44 female, 36 male), which were randomly divided into 4 groups of 20 patients each, due to the treatment type: Botulinum toxin (BTX); Dry needling (DN); Pharmacological therapy (PT) and Manual therapy (MT). All treatments were carried out by the same maxillofacial surgeon. An informed consent form was obtained from all participants.

DETAILED DESCRIPTION:
The study aimed to assess and compare the effectiveness of 4 different methods in the management bruxism: Botulinum toxin (BTX-A), dry needling (DN), pharmacological therapy (PT), and manual therapy (MT). 80 bruxist patients (44 female, 36 male) were randomly divided into 4 groups of 20 patients each. Botulinum toxin, dry needling, pharmacological therapy and manual therapy were carried out by the same maxillofacial surgeon in all patients. The following measurements were recorded by another investigator in each group, at baseline (before treatment) and at post-treatment intervals of 2nd, 4th, and 12th weeks; Visual Analogue Scale (VAS) for pain, maximum painless mouth opening (mm), Oral Health Impact Profile14 (OHIP-14).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 to 65 years with complete dentition,
* Patients classified as American Society of Anesthesiologists (ASA) physical status ASA I or ASA II
* Patients experiencing moderate to severe pain in the masticatory muscles related to bruxism,
* Patients who had not previously been treated for bruxism
* Patients who were diagnosed with bruxism were excluded from the study.

Exclusion Criteria:

* Presence of temporomandibular joint disorder
* Known allergy to botulinum toxin
* Pregnancy
* Presence of neuromuscular disease
* Chronic use of muscle relaxant medication within the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Pain in at rest and at chewing | 12 weeks
  Average pain was measured by a scale, named Visual analogue scale.
MMO | 12 weeks
  Maximum painless mouth opening (in millimeters) was measured by a special ruler.
OHRQoL questionnaire | 12 weeks
  Oral-health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: ALANUR CIFTCI SISMAN, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Sahin SS, Ciftci Sisman A, Atar E, Kilac H, Guzelce Sultanoglu E. Comparison of the effectiveness of botulinum toxin, dry needling, pharmacological treatment, and manual therapy for bruxism-induced myalgia: a prospective randomized study. J Oral Facial Pain Headache. 2024 Dec;38(4):101-110. doi: 10.22514/jofph.2024.043. Epub 2024 Dec 12. PMID 39800961